CLINICAL TRIAL: NCT00242814
Title: A Phase IV Study, Prospective, Randomised, Open Label, Blinded Endpoint, Parallel Group, 9 Weeks of Comparison Between Oral Administration of Telmisartan Tablet (80mg Once Daily) and Amlodipine Tablet (10 mg Once Daily) on Biological PPAR Gamma Activities in Non Controlled Hypertensive Male Patients With Metabolic Syndrome
Brief Title: Phase IV, 9 Weeks Comparison Between MICARDIS 80 mg and Amlodipine 10 mg on Biological PPAR Gamma Activities
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 502.486
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Hypertension; Metabolic Syndrome X
MeSH Terms: conditions — Hypertension; Metabolic Syndrome | interventions — Telmisartan; Amlodipine

INTERVENTIONS:
Drug: Micardis
Drug: Amlodipine
Procedure: Abdominal biopsy

SUMMARY:
The objective of the study is to compare PPAR activities (increase of adiponectin level) between MICARDIS and amlodipine after 6 weeks of treatment in hypertensive patients with metabolic syndrome. Moreover, this study will compare serum level of inflammatory markers of the metabolic syndrome after 6 weeks of treatment.

An ancillary study performed in one center will assess adipocyte differentiation (PPAR gamma stimulation) in 30 subjects (15 per arm).

ELIGIBILITY:
Inclusion Criteria:

Patient written informed consent is signed prior to any trial specific procedures participation

* male patients > 18 years
* Mean seated SBP > 130mmHg and/or DBP > 85mmHg treated with antihypertensive drug(s)
* with at least 2 more criteria of metabolic syndrome (NCEPT III). Biological data available within 6 months prior to enrollment visit.
* abdominal obesity > 102 cm at screening
* TG > 1.5 g/l
* HDL < 0.4 g/l
* Glycemia > 6 mmol/l

Exclusion Criteria:

Patients with any of the following conditions will be excluded from trial:

* confirmed type 1 or 2 diabetic patients treated or not
* secondary hypertension
* Mean seated SBP>180 mmHg and/or DBP >110 mmHg at screening
* hepatic and/or renal dysfunction as defined by the following laboratory parameters at visit 1:
* SGPT (ALT) or SGOT (AST) ¿ twice the upper limit of the normal range
* serum creatinine ¿ 2.3 mg/dL (or 203 ¿mol/L)
* bilateral renal artery stenosis or renal artery stenosis in a solitary kidney
* patients post-renal transplant or with only one functioning kidney
* clinically relevant hypokalemia or hyperkalemia at visit 1
* uncorrected volume or sodium depletion at visit 1
* primary aldosteronism
* hereditary or known fructose intolerance
* biliary obstructive disorders
* patients who have previously experienced symptoms characteristic of angioedema during treatment with angiotensin-II receptor antagonists
* history of drug or alcohol dependency within the previous six months
* concurrent participation in another clinical trial or any investigational therapy within thirty days prior to signing the consent form
* symptomatic congestive heart failure (New York Heart Academy (NYHA) functional class CHF II-IV)
* unstable angina pectoris, myocardial infarction, percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG) surgery less than three months prior to informed consent
* stroke less than six months prior to informed consent
* sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant arrhythmias as determined by the investigator
* hypertrophic obstructive cardiomyopathy, hemodynamically relevant stenosis of the aortic or mitral valve
* known allergic hypersensitivity to any component of the formulations under investigation
* concomitant therapy with lithium, cholestyramine or colestipol resins continued after visit 1

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-11-03 (Actual); Primary Completion 2007-03-29 (Actual)

PRIMARY OUTCOMES:
Comparison of the serum adiponectin level at the end of study (6 weeks) between the two groups. | At week 6

SECONDARY OUTCOMES:
Comparison of serum level of TNF alpha, IL-6, leptine, hsCRP, TG, HDL and blood pressure control between two groups. Adipocyte differentiation in 30 patients (PPAR gamma stimulation) between two groups. | At week 6

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (31):
- France (31):
  - 502.486.3302A Cabinet Médical, Angers
  - 502.486.3302B Cabinet Médical, Angers
  - 502.486.3303A Boehringer Ingelheim Investigational Site, Angers
  - 502.486.3305A Cabinet Médical, Angers
  - 502.486.3323A Cabinet Médical, Angers
  - 502.486.3323B Cabinet Médical, Angers
  - 502.486.3324A Cabinet Médical, Angers
  - 502.486.3324B Cabinet Médical, Angers
  - 502.486.3325A Cabinet médical, Angers
  - 502.486.3326A Cabinet Médical, Angers
  - 502.486.3328A Cabinet Médical, Angers
  - 502.486.3306A Cabinet Médical, Briollay
  - 502.486.3307A Cabinet Médical, Chemillé-Melay
  - 502.486.3319A Cabinet Médical, Cherbourg
  - 502.486.3320A Cabinet Médical, Cherbourg
  - 502.486.3320B Cabinet Médical, Cherbourg
  - 502.486.3321A Cabinet Médical, Équeurdreville-Hainneville
  - 502.486.3322A Boehringer Ingelheim Investigational Site, Évron
  - 502.486.3312A Cabinet Médical, Feneu
  - 502.486.3315A Cabinet Médical, La Rochelle
  - 502.486.3308A Cabinet Médical, Montrevault
  - 502.486.3316A Boehringer Ingelheim Investigational Site, Nieul-sur-Mer
  - 502.486 3301A Boehringer Ingelheim Investigational Site, Paris
  - 502.486.3301B Hôpital Pitié Salpêtrière, Paris
  - 502.486.3310A Cabinet Médical, Saint-Pierre-Montlimart
  - 502.486.3327A Cabinet Médical, Saumur
  - 502.486.3309A Cabinet Médical Jean Charcot, Segré
  - 502.486.3311A Cabinet Médical, Tiercé
  - 502.486.3311B Cabinet Médical, Tiercé
  - 502.486.3311C Cabinet Médical, Tiercé
  - 502.486.3311D Cabinet Médical, Tiercé